CLINICAL TRIAL: NCT06557460
Title: A Phase IIb, Randomized, Assessor-Masked, Multicenter Clinical Trial to Assess the Safety and Efficacy of Subretinal Implantation of the CPCB-RPE1 Implant in Subjects With Advanced, Dry Age-Related Macular Degeneration (Geographic Atrophy) - PATCH AMD
Brief Title: A Phase IIb Randomized, Multicenter Trial of Subretinal CPCB-RPE1 in Advanced Dry AMD (Geographic Atrophy)
Acronym: PATCH-AMD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regenerative Patch Technologies, LLC (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RPT-14-02
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Dry Age-related Macular Degeneration; Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: Phase IIb, Randomized, Assessor-Masked, Multicenter Clinical Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active treatment group receiving the CPCB-RPE1 implant (up to 18 subjects). (Experimental): Active treatment group receiving the CPCB-RPE1 implant (up to 18 subjects).
  Interventions: Device: Surgical implantation of the CPCB-RPE1 implant
- Control group receiving a simulated "sham" implantation procedure (up to 6 subjects) (Sham Comparator): Control group receiving a simulated "sham" implantation procedure (up to 6 subjects)
  Interventions: Device: Surgical implantation of the CPCB-RPE1 implant

INTERVENTIONS:
Device: Surgical implantation of the CPCB-RPE1 implant — Surgical implantation of the CPCB-RPE1 implant

SUMMARY:
This is a Phase IIb randomized, clinical trial designed to assess the safety and efficacy of unilateral implantation of the CPCB-RPE1 implant in subjects with geographic atrophy involving the fovea.

Up to 6 surgical implantation sites will deliver the CPCB-RPE1 in this Phase IIb clinical trial. Additional study sites may serve as referral or follow-up sites. Twenty-four (24) subjects will participate in the trial and will be randomized 3:1 to one of 2 groups:

* The treatment group receiving the CPCB-RPE1 implant (up to 18 subjects).
* The control group receiving a simulated "sham" implantation procedure (up to 6 subjects)

ELIGIBILITY:
Eligible participants include:

1. Age 55 to 90 years of age (inclusive), presenting with geographic atrophy involving the fovea in advanced, age-related, dry AMD.
2. Clinical findings consistent with advanced dry AMD with evidence of one or more areas of ≥4.0mm2 but not exceeding 15.0 mm2 of geographic atrophy involving the fovea.
3. Geographic atrophy defined as attenuation or loss of RPE as observed by biomicroscopy, OCT, or FAF.
4. The best-corrected visual acuity (BCVA) of the eye to receive the implant will be ≥20/200 (35 EDTRS letters) to 20/63 (60 EDTRS letters) inclusive. The BCVA of the eye that is NOT to receive the implant will be better or equal to the eye that will receive the implant.
5. Medically suitable to undergo pars plana vitrectomy and the surgical implant procedure, including being able to position post-operatively and use post-operative medications as required.
6. Medically suitable for general anesthesia or monitored intravenous sedation, if needed.
7. Pseudophakic in the study eye, to remove the risk of cataract formation following vitrectomy.
8. Participants also must be willing and able to provide written, signed informed consent for this study.
9. Participants able to complete the baseline microperimetry retinal sensitivity testing.
10. On baseline microperimetry, participants must have ≥5 spots in the perilesional region with a retinal sensitivity between 3 and 17 Db.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Change in retinal sensitivity | 1 year post implantation
  Change in retinal sensitivity by microperimetry

SECONDARY OUTCOMES:
Change in best corrected visual acuity | 1 year post implantation
  Change in best corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Associates of Southern California, Huntington Beach, California
  - USC - Keck, Los Angeles, California
  - University Retina, Lemont, Illinois
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No